CLINICAL TRIAL: NCT02105324
Title: The Summer Camp Study 2: Outpatient Automated Blood Glucose Control With a Bi-Hormonal Bionic Endocrine Pancreas in a Pediatric Population Ages 6-11 at the Clara Barton Diabetes Camps
Brief Title: The Summer Camp Study 2: Blood Glucose Control With a Bi-Hormonal Endocrine Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000630
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Type 1 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; continuous glucose monitoring (CGM); outpatient; insulin pump; pediatrics; children; camp; summer camp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Muscle Cramp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bionic Pancreas (Experimental): Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 5 days.
  Interventions: Device: Bionic Pancreas
- Usual Care (Experimental): Usual Care diabetes management in a diabetes camp environment including a nurse or nursing student assigned to each cabin and review and adjustment of the insulin regimen daily by a physician or nurse practitioner, all participants using the participant's own insulin pump and a continuous glucose monitor if they use one as part of their usual care, for 5 days.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Bionic Pancreas — Automated blood glucose control via a closed-loop bionic pancreas device.
  Other Names: Boston University Bionic Pancreas
  Arms: Bionic Pancreas
Other: Usual Care — As a comparator control, usual diabetes camp care with the participant's own insulin pump.
  Arms: Usual Care

SUMMARY:
This study will test the hypothesis that a wearable automated bionic pancreas system that automatically delivers both insulin and glucagon can improve glycemic control vs. usual care for young people with type 1 diabetes ages 6-11 years old in a diabetes camp environment.

ELIGIBILITY:
Inclusion Criteria

* Age 6-11 years with type 1 diabetes for at least one year
* Diabetes managed using an insulin infusion pump for ≥ three months
* Willing to wear two infusion sets and continuous glucose monitoring (CGM) sensor and change sets frequently (at least one new glucagon infusion set daily)
* Otherwise healthy (mild chronic disease such as asthma will be allowed if well controlled that do not require medications that result in exclusion)

Exclusion Criteria

* Unable to provide informed consent, informed assent or parental consent
* Unable to comply with study procedures
* Current participation in another diabetes-related clinical trial that, in the judgment of the principal investigator, will compromise the results of this study or the safety of the subject
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis)
* Pregnancy (positive urine human chorionic gonadotropin [HCG])
* History of liver disease that is expected to interfere with the anti-hypoglycemia action of glucagon (e.g. liver failure or cirrhosis). Other liver disease (i.e. active hepatitis, steatosis, active biliary disease, any tumor of the liver, hemochromatosis, glycogen storage disease) may exclude the subject if it causes significant compromise to liver function or may do so in an unpredictable fashion
* Personal history of cystic fibrosis, pancreatitis, or other pancreatic disease, including pancreatic tumor or insulinoma
* History of prolonged QT or arrhythmia, congenital heart disease or current known cardiac disease
* Acute illness (other than non-vomiting viral illness) or exacerbation of chronic illness other than type 1 diabetes (T1D) at the time of the study
* Seizure disorder, history of any seizure within the last two years, or ongoing treatment with anticonvulsants
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with second generation anti-psychotic medications, which are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to radio-frequency (RF) interference
* Use of oral (e.g. thiazolidinediones, biguanides, sulfonylureas, glitinides, dipeptidyl peptidase 4 (DPP-4) inhibitors, sodium-glucose linked transporter 2 (SGLT-2) inhibitors) anti-diabetic medications
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Unwilling or unable to completely avoid acetaminophen during the comparator and bionic pancreas arms of the study
* History of eating disorder such as anorexia, bulimia, or diabulemia or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Any factors that, in the opinion of the principal investigator, would interfere with the safe completion of the study procedures

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Russell SJ, Hillard MA, Balliro C, Magyar KL, Selagamsetty R, Sinha M, Grennan K, Mondesir D, Ekhlaspour L, Zheng H, Damiano ER, El-Khatib FH. Day and night glycaemic control with a bionic pancreas versus conventional insulin pump therapy in preadolescent children with type 1 diabetes: a randomised crossover trial. Lancet Diabetes Endocrinol. 2016 Mar;4(3):233-243. doi: 10.1016/S2213-8587(15)00489-1. Epub 2016 Feb 3. PMID 26850709
- See also: Information about this and related studies — http://www.bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Bionic Pancreas Then Usual Care: Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 5 days in Period 1, followed by Usual Care diabetes management in a diabetes camp environment including a nurse or nursing student assigned to each cabin and review and adjustment of the insulin regimen daily by a physician or nurse practitioner, all participants using the participant's own insulin pump and a continuous glucose monitor if they use one as part of their usual care, for 5 days in Period 2. There was a 3-day washout period between periods.
- Usual Care Then Bionic Pancreas: Usual Care diabetes management in a diabetes camp environment including a nurse or nursing student assigned to each cabin and review and adjustment of the insulin regimen daily by a physician or nurse practitioner, all participants using the participant's own insulin pump and a continuous glucose monitor if they use one as part of their usual care, for 5 days in Period 1, followed by Bionic Pancreas diabetes management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a CGM device, for 5 days in Period 2. There was a 3-day washout period between periods.
Period: Period 1
Arm/Group | Bionic Pancreas Then Usual Care | Usual Care Then Bionic Pancreas
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Bionic Pancreas Then Usual Care | Usual Care Then Bionic Pancreas
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who completed both periods of the study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Continuous Glucose Monitoring Glucose (CGMG) Values During Days 2 to 5
Description: Glucose reading were taken every 5 minutes by the CGM. The CGM glucose results during Days 2 through 5 were averaged.
Time Frame: Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
milligrams/deciliter (mg/dL) | 136.8 (10.8) | 167.4 (30.6)

2. Primary Outcome: Percentage of Time Spent With CGMG Concentration < 60 mg/dL During Days 2 to 5
Description: Glucose reading were taken every 5 minutes by the CGM. The percentage of time that the glucose concentration was less than 60 mg/dL [3.3 millimoles/liter (mmol/L)] during Days 2 through 5 was calculated.
Time Frame: Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time | 1.2 (1.1) | 2.8 (1.2)

3. Secondary Outcome: Mean CGMG Values
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose results for each time frame were averaged.
Time Frame: Day 1 and Days 1-5 in each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
mg/dL
  Day 1 | 153.6 (19.7) | 179.2 (37.8)
  Days 1 to 5 | 140.6 (12.0) | 169.9 (27.6)

4. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Day 1
Description: Glucose readings were taken every 5 minutes by the CGM. The percentage of time that the glucose concentration was less than the following ranges were calculated: < 50 mg/dL(2.8 mmol/L), < 70 mg/dL (3.9 mmol/L), 70-180 mg/dL (3.9 to 10.0 mmol/L), > 180 mg/dL (10.0 mmol/L).
Time Frame: Day 1 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time
  < 50 mg/dL (2.8 mmol/L) | 0.2 (0.6) | 1.0 (2.6)
  < 70 mg/dL (3.9 mmol/L) | 1.8 (2.0) | 3.7 (4.5)
  70-180 mg/dL (3.9 to 10.0 mmol/L) | 71.6 (11.7) | 52.1 (21.3)
  > 180 mg/dL (10.0 mmol/L) | 26.6 (11.3) | 44.2 (23.4)

5. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Days 1 to 5
Description: Glucose readings were taken every 5 minutes by the CGM. The percentage of time that the glucose concentration was less than the following ranges were calculated: < 50 mg/dl (2.8 mmol/L), < 70 mg/dl (3.9 mmol/L), 70-180 mg/dl (3.9 to 10.0 mmol/L), > 180 mg/dL (10.0 mmol/L).
Time Frame: Days 1 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time
  < 50 mg/dl (2.8 mmol/L) | 0.4 (0.4) | 1.1 (0.8)
  < 70 mg/dl (3.9 mmol/L) | 2.7 (1.8) | 5.6 (2.5)
  70-180 mg/dl (3.9 to 10.0 mmol/L) | 78.8 (7.4) | 56.5 (13.9)
  > 180 mg/dL (10.0 mmol/L) | 18.5 (6.6) | 37.9 (15.4)

6. Secondary Outcome: Percentage of Time With CGMG Concentration by Ranges During Days 2 to 5
Description: as for outcome 5
Time Frame: Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time
  < 50 mg/dl (2.8 mmol/L) | 0.4 (0.5) | 1.1 (0.8)
  < 70 mg/dl (3.9 mmol/L) | 2.9 (2.1) | 6.1 (2.8)
  70-180 mg/dl (3.9 to 10.0 mmol/L) | 80.6 (7.4) | 57.6 (14.0)
  > 180 mg/dL (10.0 mmol/L) | 16.5 (6.4) | 36.3 (15.7)

7. Secondary Outcome: Percentage of Participants With Mean CGMG Glucose <154 mg/dL
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose readings were averaged. 154 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 7.0%.
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 57.9 | 15.8
  Days 1 to 5 | 84.2 | 36.8
  Days 2 to 5 | 94.7 | 42.1

8. Secondary Outcome: Percentage of Participants With Mean CGMG Glucose <169 mg/dL
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose readings were averaged. 169 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 7.5%.
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 89.5 | 36.8
  Days 1 to 5 | 94.7 | 57.9
  Days 2 to 5 | 100 | 68.4

9. Secondary Outcome: Percentage of Participants With Mean CGMG Glucose <183 mg/dL
Description: Glucose reading were taken every 5 minutes by the CGM. The glucose readings were averaged. 183 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 8.0%.
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 89.5 | 57.9
  Days 1 to 5 | 100 | 68.4
  Days 2 to 5 | 100 | 73.7

10. Secondary Outcome: Number of CGMG Reported Hypoglycemic Events (< 70 mg/dL, < 60 mg/dL, <50 mg/dL)
Description: A series of hypoglycemic measurements is defined as a single event until there is a break of ≥ 30 minutes between measurements below the defined thresholds of < 70, < 60, and <50 mg/dL.
Time Frame: Days 1-5
Measure: Mean (Standard Deviation); unit: times below threshold
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
times below threshold
  <70 mg/dl | 9.4 (5.8) | 9.4 (5.1)
  <60 mg/dl | 4.4 (3.3) | 6.3 (3.0)
  <50 mg/dl | 1.9 (1.9) | 3.1 (2.1)

11. Secondary Outcome: Mean Plasma Glucose Values
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). The plasma glucose readings were averaged. The plasma glucose results on Day 1, Days 1 to 5 and Days 2 to 5 were averaged.
Time Frame: Day 1, Days 1 to 5, and Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
mg/dL
  Day 1 | 137.2 (20.1) | 169.7 (32.2)
  Days 1 to 5 | 136.8 (7.2) | 176.4 (25.2)
  Days 2 to 5 | 135.8 (5.4) | 178.8 (27.4)

12. Secondary Outcome: Percentage of Time With Plasma Glucose Values by Ranges on Day 1
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). The percentage of time that the plasma glucose concentration was less than the following ranges were calculated: < 70 mg/dl (3.9 mmol/L), < 60 mg/dL (3.3 mmol/L), < 50 mg/dl (2.8 mmol/L).
Time Frame: Day 1 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of values
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of values
  < 70 mg/dL (3.9 mmol/L) | 4.4 (0.1) | 3.7 (0.07)
  < 60 mg/dL (3.3 mmol/L) | 0.9 (0.4) | 2.8 (0.06)
  < 50 mg/dL (2.8 mmol/L) | 0 (0) | 0.9 (0.04)

13. Secondary Outcome: Percentage of Time With Plasma Glucose Values by Ranges on Days 1 to 5
Description: as for outcome 12
Time Frame: Days 1 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of values
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of values
  < 70 mg/dL (3.9 mmol/L) | 2.7 (0.03) | 4.3 (0.04)
  < 60 mg/dL (3.3 mmol/L) | 1.1 (0.02) | 2.1 (0.02)
  < 50 mg/dL (2.8 mmol/L) | 0.4 (0.01) | 0.5 (0.01)

14. Secondary Outcome: Percentage of Time With Plasma Glucose Values by Ranges on Days 2 to 5
Description: as for outcome 12
Time Frame: Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of values
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of values
  < 70 mg/dl (3.9 mmol/L) | 2.2 (0.03) | 4.4 (0.04)
  < 60 mg/dL (3.3 mmol/L) | 1.1 (0.02) | 1.9 (0.02)
  < 50 mg/dl (2.8 mmol/L) | 0.4 (0.013) | 0.2 (0.01)

15. Secondary Outcome: Percentage of Participants With Mean Plasma Glucose <154 mg/dL
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). The plasma glucose readings were averaged. 154 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 7.0%.
Time Frame: Day 1, Days 1 to 5, and Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 84 | 37
  Days 1 to 5 | 100 | 16
  Days 2 to 5 | 100 | 11

16. Secondary Outcome: Percentage of Participants With Mean Plasma Glucose <169 mg/dL
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). The plasma glucose readings were averaged. 169 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 7.5%.
Time Frame: Day 1, Days 1 to 5, and Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 95 | 58
  Days 1 to 5 | 100 | 37
  Days 2 to 5 | 100 | 53

17. Secondary Outcome: Percentage of Participants With Mean Plasma Glucose <183 mg/dL
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). The plasma glucose readings were averaged. 183 mg/dL was the estimated average glucose corresponding to a Hemoglobin A1C of 8.0%.
Time Frame: Day 1, Days 1 to 5, and Days 2 to 5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of participants
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of participants
  Day 1 | 95 | 68
  Days 1 to 5 | 100 | 68
  Days 2 to 5 | 100 | 63

18. Secondary Outcome: Number of Plasma Glucose Reported Hypoglycemic Events (< 70 mg/dL, < 60 mg/dL, <50 mg/dL)
Description: as for outcome 10
Time Frame: Days 1-5
Measure: Mean (Standard Deviation); unit: times below threshold
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
times below threshold
  <50 mg/dl | 0.47 (0.61) | 0.53 (0.61)
  <60 mg/dl | 1.26 (1.19) | 2.11 (1.97)
  <70 mg/dl | 2.84 (2.39) | 4.79 (3.52)

19. Secondary Outcome: Percentage of Days That CGM Data Was Used by Participants as Part of Their Usual Care
Description: The percentage of days during the Usual Care period that participants used CGM data as part of their diabetes management.
Time Frame: Day 1, Days 1-5, and Days 2-5 of the Usual Care Period
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: percentage of days
Arm/Group | Usual Care
Number analyzed (Participants) | 19
percentage of days
  Day 1 | 0
  Days 1 to 5 | 0
  Days 2 to 5 | 0

20. Secondary Outcome: Number of Carbohydrate Interventions for Hypoglycemia When Plasma Glucose <70 mg/dL
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). Participants were given 15 grams (g) of simple carbohydrates if their plasma glucose concentration dropped below 4.4 mmol/L. These simple carbohydrates were counted as interventions for study outcomes if the plasma glucose concentration was less than 3.9 mmol/L. A second intervention of 15 g of carbohydrate was given if a repeat measurement in 15-20 min was less than 3.9 mmol/L. The total number of carbohydrate interventions are reported.
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Median (Full Range); unit: carbohydrate interventions
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
carbohydrate interventions
  Day 1 | 1 [0 to 3] | 1 [0 to 5]
  Days 1 to 5 | 3 [0 to 8] | 5 [0 to 14]
  Days 2 to 5 | 2 [0 to 7] | 3 [0 to 11]

21. Secondary Outcome: Grams of Carbohydrate Taken for Hypoglycemia When Plasma Glucose <70 mg/dL
Description: Fingerstick plasma glucose measurements were obtained before meals, at bedtime, at midnight, and at about 3:45 AM (six scheduled measurements). Participants were given 15 grams (g) of simple carbohydrates if their plasma glucose concentration dropped below 4.4 mmol/L. These simple carbohydrates were counted as interventions for study outcomes if the plasma glucose concentration was less than 3.9 mmol/L. A second intervention of 15 g of carbohydrate was given if a repeat measurement in 15-20 min was less than 3.9 mmol/L.
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All randomized participants who completed both periods of the study.
Measure: Median (Full Range); unit: grams of carbohydrate
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
grams of carbohydrate
  Day 1 | 1.6 [0 to 8] | 2.2 [0 to 10]
  Days 1 to 5 | 7.3 [0 to 19] | 12.7 [0 to 40]
  Days 2 to 5 | 5.7 [0 to 16] | 9.6 [0 to 31]

22. Secondary Outcome: Insulin Total Daily Dose
Description: Insulin total daily dose is reported in units per kilogram per day (U/kg/day).
Time Frame: 11 days
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
U/kg/day
  Day 1 | 0.7 (0.2) | 0.66 (0.15)
  Days 1 to 5 | 0.68 (0.14) | 0.68 (0.13)
  Days 2 to 5 | 0.68 (0.15) | 0.68 (0.13)

23. Secondary Outcome: Glucagon Total Daily Dose Levels in the Bionic Pancreas Arm
Description: Glucagon dose level is reported in micrograms per kilogram of body mass per day (µg/kg/day).
Time Frame: Day 1, Days 1-5, and Days 2-5 of each period
Population: All participants who completed both periods of the study. Results are reported for the Bionic Pancreas period only.
Measure: Mean (Standard Deviation); unit: µg/kg/day
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 19
µg/kg/day
  Day 1 | 11.9 (5.2)
  Days 1 to 5 | 11.1 (3.8)
  Days 2 to 5 | 10.9 (4.0)

24. Secondary Outcome: Daily Basal Insulin Dose in the Bionic Pancreas Period
Description: The bionic pancreas automatically adapted insulin dosing to each individual's needs. When CGM data were not available (because of sensor failure or during the warm-up time after sensor replacement), the bionic pancreas automatically delivered a dose of basal insulin based on the mean basal dosing it had calculated at that time on previous days. Daily basal insulin dose is reported in units per kilogram (kg) per day (U/kg).
Time Frame: Day 1 through Day 5
Population: All participants who completed both periods of the study. Results are reported for the Bionic Pancreas period only.
Measure: Mean (Standard Deviation); unit: U/kg/day
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 19
U/kg/day
  Day 1 | 0.2 (0.0)
  Day 2 | 0.3 (0.1)
  Day 3 | 0.3 (0.1)
  Day 4 | 0.3 (0.0)
  Day 5 | 0.3 (0.1)

25. Secondary Outcome: Daily Bolus Insulin Dose in the Bionic Pancreas Period
Description: The first time the bionic pancreas was used in each participant, a partial meal-priming bolus based on the participant's body mass (0.05 units/kg) was delivered. After the first use, the size of the meal-priming bolus was adapted by the bionic pancreas to 75% of the 4-hour prandial insulin used for that meal type and size. Daily bolus insulin dose is reported in units per kilogram (kg) per day (U/kg).
Time Frame: Day 1 through Day 5
Population: All participants who completed both periods of the study. Results are reported for the Bionic Pancreas period only.
Measure: Mean (Standard Deviation); unit: U/kg/day
Groups:
- Bionic Pancreas: Participants who were randomized and began in the trial
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 19
U/kg/day
  Day 1 | 0.4 (0.1)
  Day 2 | 0.4 (0.2)
  Day 3 | 0.4 (0.1)
  Day 4 | 0.4 (0.1)
  Day 5 | 0.4 (0.1)

26. Secondary Outcome: Carbohydrate Intake
Description: Carbohydrate intake included meals, snacks and unscheduled carbohydrates administered when a participant's blood glucose was <80 mg/dl (or for symptoms at any glucose level). Carbohydrate intake per day was averaged and is reported in grams (g) per kilogram (kg) per day (g/kg/day).
Time Frame: Day 1, Days 1-5 and Days 2-5
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: g/kg/day
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
g/kg/day
  Day 1 | 5.51 (1.46) | 6.09 (2.08)
  Days 1 to 5 | 6.09 (1.53) | 6.66 (1.72)
  Days 2 to 5 | 6.24 (1.62) | 6.80 (1.70)

27. Secondary Outcome: Number of Unscheduled Infusion Set Changes
Description: Infusion sets for administering insulin and glucagon were placed under the skin the in the abdomen, buttocks, arms, or legs. Infusion set changes due to pain, infusion set falling out or infusion set failure are reported. Camp policy was to suspect failure of the infusion set whenever ketonemia occurred, so failures may not have actually been set failures, but rather failure to deliver enough insulin.
Time Frame: Day 1
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: unscheduled infusion set changes
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
unscheduled infusion set changes
  Fell out | 1 | 0
  Failure | 0 | 1
  Pain | 1 | 0

28. Secondary Outcome: Number of Unscheduled Infusion Set Changes
Description: as for outcome 27
Time Frame: Days 1-5
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: unscheduled infusion set changes
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
unscheduled infusion set changes
  Fell out | 7 | 1
  Failure | 2 | 5
  Pain | 3 | 0

29. Secondary Outcome: Number of Unscheduled Infusion Set Changes
Description: as for outcome 27
Time Frame: Days 2-5
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: unscheduled infusion set changes
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
unscheduled infusion set changes
  Fell out | 6 | 1
  Failure | 2 | 4
  Pain | 2 | 0

30. Secondary Outcome: Number of Bionic Pancreas Local Infusion Site Reactions
Description: Local infusion site reactions are defined as pain at the infusion site of the Bionic Pancreas. Itching and redness may have also been present.
Time Frame: Day 1, Days 1-5 and Days 2-5
Population: All randomized participants who completed both periods of the study. Results are reported for the Bionic Pancreas period only.
Measure: Number; unit: infusion site reactions
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 19
infusion site reactions
  Day 1 | 1
  Days 1 to 5 | 3
  Days 2 to 5 | 2

31. Secondary Outcome: Mean Nausea Index Score Using a Visual Analogue Scale (VAS)
Description: Participants rated their nausea using a 0 to 10 centimeter (cm) VAS where 0=least severe nausea to 10=most severe nausea. The average nausea index scores from Day 1 to Day 5 were calculated
Time Frame: Day 1, Days 1-5, and Days 2-5 in each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
cm
  Day 1 | 1.1 (2.2) | 0.9 (2.2)
  Days 1 to 5 | 1.3 (2.0) | 1.4 (1.8)
  Days 2 to 5 | 1.4 (2.3) | 1.5 (1.8)

32. Secondary Outcome: Number of Severe Hypoglycemic Events
Description: A severe hypoglycemic event is an event where the participant is unable to self-treat and requires the assistance of another person.
Time Frame: Day 1, Days 1-5 and Days 2-5
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: severe hypoglycemic events
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
severe hypoglycemic events
  Day 1 | 0 | 0
  Days 1 to 5 | 0 | 0
  Days 2 to 5 | 0 | 0

33. Secondary Outcome: Percentage of Time Participants Were Not Under Bionic Pancreas Control During the Bionic Pancreas Period
Description: Percentage of time that the Bionic pancreas was not functioning properly due to loss of wireless connectivity.
Time Frame: 5 days
Population: All randomized participants who completed both periods of the study. Reported for the Bionic Pancreas period only.
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Bionic Pancreas: management, a wearable bionic pancreas system that automatically delivers insulin and glucagon using a continuous glucose monitoring (CGM) device, for 5 days.
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 19
percentage of time
  Insulin Pump: Loss of Wireless Connectivity | 4.9 (2.5)
  Glucagon Pump: Loss of Wireless Connectivity | 6.1 (3.1)

34. Secondary Outcome: Percentage of Time Without CGM Monitoring Data
Description: Percentage of time without CGM monitoring data is the time when the participant's CGM device lost its CGM signal.
Time Frame: 5 days
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time | 4.2 (1.9) | 5.1 (1.9)

35. Secondary Outcome: Change From Baseline in Body Weight
Description: The change in body weight collected at Day 5 of each period relative to Baseline. A negative change from Baseline indicates a reduction in body weight and a positive change from Baseline indicates an increase in body weight.
Time Frame: 5 days
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
kg | 0.07 (0.63) | 0.28 (0.81)

36. Secondary Outcome: Reliability Index
Description: Reliability index was calculated as the percentage of time values were actually recorded by CGM.
Time Frame: Day 1, Days 1-5, and Days 2-5 in each period
Population: All randomized participants who completed both periods of the study.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
percentage of time
  Day 1 | 95.3 (3.76) | 95.1 (2.28)
  Days 1 to 5 | 95.4 (2.0) | 93.1 (3.0)
  Days 2 to 5 | 95.8 (1.9) | 95.0 (1.9)

37. Secondary Outcome: List of Technical Faults Associated With the Bionic Pancreas Including Cause and Resolution
Time Frame: 5 days
Population: Data was not collected and analyzed to this level of detail.
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Number of Unscheduled CGM Sensor Changes
Description: The number of time a CGM sensor was replaced due to falling out or failing to report a glucose value.
Time Frame: 5 days
Population: All randomized participants who completed both periods of the study.
Measure: Number; unit: CGM sensor changes
Arm/Group | Bionic Pancreas | Usual Care
Number analyzed (Participants) | 19 | 19
CGM sensor changes | 3 | 5

39. Secondary Outcome: Percentage of Participants Using a Glucagon-Like Peptide-1 (GLP-1) Agonist During the Usual Care Period
Description: The percentage of participants who used a GLP-1 agonist to manage their diabetes during the Usual Care period.
Time Frame: 5 days
Population: All participants who completed both periods of the study. Results are reported for the Usual Care period only.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care
Number analyzed (Participants) | 19
percentage of participants | 0

40. Secondary Outcome: Percentage of Participants Using Pramlintide During the Usual Care Period
Description: The percentage of participants who used pramlintide to manage their diabetes during the Usual Care period.
Time Frame: 5 days
Population: All participants who completed both periods of the study. Results are reported for the Usual Care period only.
Measure: Number; unit: percentage of participants
Arm/Group | Usual Care
Number analyzed (Participants) | 19
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 5 days for each arm
Arm/Group | Bionic Pancreas | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 15/19 | 13/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bionic Pancreas (N=19) | Usual Care (N=19)
Hyperketonemia (Investigations) | 0 | 5
Vomiting in mouth (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Stomachache (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 14 | 11
Infusion site pain (General disorders) | 3 | 0
Infusion site redness (General disorders) | 2 | 0
Infusion site itching (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No